CLINICAL TRIAL: NCT00229242
Title: Comparison of Diuretic-based With Non-diuretic Based Hypertension Therapy Using Echocardiographic Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Dr Kofo Ogunyankin, Queens University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DMED-676-03
Record Dates: First submitted 2005-09-13; First posted 2005-09-29 (Estimated); Last update posted 2009-12-14 (Estimated); Status verified 2009-12

CONDITIONS: Hypertension
Keywords: Ambulatory blood pressure monitoring; Echocardiography; Diastolic function; Left ventricular mass regression
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Diuretic-Based Hypertension Therapy
  Interventions: Drug: Diuretic-Based or Non-Diuretic Based Hypertension Therapy
- 2 (Active Comparator): Non-Diuretic-Based Hypertension Therapy
  Interventions: Drug: Diuretic-Based or Non-Diuretic Based Hypertension Therapy

INTERVENTIONS:
Drug: Diuretic-Based or Non-Diuretic Based Hypertension Therapy

SUMMARY:
MAIN: The benefits of treating high blood pressure successfully to normal levels on heart function are the same regardless of which particular combination of drugs are used. SECONDARY: Measurement of heart function using a comprehensive ultrasound imaging method (Echocardiography) and an objective test of functional ability are better predictors of changes in heart function with successful hypertension treatment, than subjective signs of heart failure.

DETAILED DESCRIPTION:
Successful treatment of hypertension with single medications is very rare. On average successful treatment requires more than 2 medications. These medications work by different methods. One of the ideas behind the use of combinations of medication for hypertension is that benefits are additive. There are unresolved questions about whether the observed benefits are simply related to effective treatment of hypertension, or whether some of the medications have special benefits independent of blood pressure lowering. Each of these contentions has been justified by clinical trials. However these trials have in common the flaw that hypertension is either not effectively controlled in all the treated subjects, or the magnitude of blood pressure change after treatment is different in the groups compared. The result of one of the largest blood pressure clinical trials called ALLHAT trial has recently fuelled this debate. The ALLHAT trial which utilized only subjective symptoms and signs of heart failure, called the FRAMINGHAM score, to determine who has abnormal heart function, implied that diuretics (water pills) were superior to the newer drugs in reducing the frequency of abnormal heart function. This study shared the flaw of previous trials in not having equal blood pressure lowering in the groups. Nevertheless it provided some evidence that argued against the notion that newer drugs were better than older drugs like diuretics. Shortly after the publication of ALLHAT, another trial called ANBP was published showing that the group of drugs that was least effective in ALLHAT was superior to diuretics in preventing important cardiovascular outcomes. Hence, it is not currently clear that there are differences between various drug combinations, if effective and equal blood pressure lowering is achieved. Another finding that may have confounded clinical trials that rely on subjective scores of heart dysfunction such as the ALLHAT, is that a significant proportion of subjects with advanced heart disease are unaware of their heart problem and hence will probably not seek attention. This raises the concern that the true frequency of abnormal heart function might not have been reported in those studies. Using more modern tools such as Echocardiography, a more complete assessment of heart dysfunction can be obtained. In addition objective tests of heart function such as the 6-minute walk distance could yield a more reliable assessment of any worsening or improvement in heart function if performed serially in treated subjects. In view of the above discussion, only a study in which hypertension is effectively and similarly controlled could be used to answer the questions regarding different effects of various drug combinations. Such is this study proposed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-65 years;
2. Hypertension with average 24-hour BP of >130 mmHg systolic or >80 mmHg diastolic in spite of treatment with one medication;
3. Office systolic blood pressure >140 mmHg and less than 180mmHg;
4. Able to comprehend and sign the consent form;
5. Able to tolerate either hydrochlorothiazide 25 mg or amlodipine 5 mg daily for 3 weeks during the run-in phase.

Exclusion Criteria:

1. Diagnosis of secondary hypertension;
2. Hypertension with systolic BP >180 mmHg in spite of 1 medication;
3. Chronic heart failure requiring diuretics, Angina or coronary syndrome requiring anti-angina therapy with CCB or beta blockers, or more than 0.4 mg/hr nitroglycerine patch;
4. Left Ventricular Ejection Fraction (LVEF) <20% or LV end systolic dimension >75 mm;
5. Significant valvular disease such as; more than mild disease of aortic or mitral valve;
6. Technically sub-optimal acoustic window or regional wall motion abnormalities;
7. Patients currently on both CCB and diuretics for more than 4 weeks;
8. Normal 24 hour ABPM at the end of the run-in period;
9. Physical handicap that precludes adequate performance of 6-minute walk such as arthritis;
10. Concomitant comorbidity that might compromise ability to evaluate treatment or enhance risks of therapy, such as: atrial fibrillation with resting ventricular rate of >100 bpm; morbid obesity; uncontrolled diabetes mellitus; severe chronic obstructive pulmonary disease (COPD); hypertrophic cardiomyopathy; and documented history of non-compliance with treatment;
11. Any condition or disorder other than hypertension that: Requires prolonged hospitalization; May limit life expectancy within 2 years; would increase the risk of participation to the subject (in the opinion of the investigator).

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-11; Primary Completion 2006-12 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Measurement of systolic and diastolic function in responders to therapy | 0, 3 and 6 months
LV mass in responders | 0, 3 and 6 months
Change in 6-minute walk distance in responders | 0, 3, and 6 months

SECONDARY OUTCOMES:
Correlation between interval improvement or deterioration in Framingham score and corresponding change in echocardiographic classification in all subjects | 3 and 6 months
Correlation between interval improvement or deterioration in LV Mass and corresponding change in 6 minute walk distance and diastolic function in all subjects | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kofo O Ogunyankin, MD, FACC, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Result] Ogunyankin KO, Day AG. Successful treatment of hypertension accounts for improvements in markers of diastolic function - a pilot study comparing hydrochlorothiazide-based and amlodipine-based treatment strategies. Can J Cardiol. 2009 Dec;25(12):e406-12. doi: 10.1016/s0828-282x(09)70534-3. PMID 19960134